CLINICAL TRIAL: NCT06669273
Title: Oncological Prognosis of Prostate Lesions by CEST MRI: Correlation of CEST MRI and Anatomopathological Analysis
Brief Title: Oncological Prognosis of Prostate Lesions by Chemical Exchange Saturation Transfer Magnetic Resonance Imaging (CEST-MRI)
Acronym: ProstaCEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2024 CHABROT; 2024-A01950-47 (Other: ANSM)
Record Dates: First submitted 2024-10-21; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Suspected Prostate Cancer (increased PSA Level)
Keywords: suspected prostate cancer; increased PSA level; CEST-MRI; Guanidyl/APT ratio to assess tumor acidosis,; tumor classification; Gleason score; PI-RADS score

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 : - Label : suspicion of prostate cancer (Experimental): Patients will be included:
  * aged over 18
  * with suspected prostate cancer identified by an increase in blood PSA concentration
  * naïve to chemotherapy, radiotherapy or hormonal therapy
  * affiliated to a Social Security system
  * able to give informed consent to participate in research
  * understanding and reading French well
  Interventions: Other: CEST MRI sequence at 3T

INTERVENTIONS:
Other: CEST MRI sequence at 3T — The MRI will be performed at the Clermont Ferrand University Hospital on the 3T research MRI on a Siemens MRI system (MAGNETOM VIDA, Siemens Healthcare, Erlangen, Germany), the emission of the radiofrequency pulses and the reception of the signal will be done using a coil dedicated to the abdo-pelvic region. The images will be analyzed by the radiologist.
  MRI is non-irradiating medical imaging. It is practiced according to good practices and the recommendations of the French Society of Radiology.
  * Acquisition of morphological T1, T2 sequences for the identification of areas of interest on the pelvic area.
  * Acquisition of the CEST MRI sequence (acquisition time 5 min)
  * Acquisition of functional sequences, DWI diffusion-weighted images and dynamic DCE sequence after injection of a single dose of non-linear gadolinum.
  The imaging report will reveal the presence or absence of tumor lesions in the prostate and their location. Data will then be compared to the histopathological analysis.

SUMMARY:
Prostate cancer is the second most common type of cancer in men only after lung cancer, and accounts for ~3.8% of all deaths caused in men in 2018. Multiparametric MRI, which combines anatomical MRI sequences (T2-weighted acquisitions) and functional sequences (DWI Diffusion-Weighted Imaging or dynamic contrast-enhanced (DCE) acquisitions), constitutes a key tool in the detection and monitoring of the therapeutic response in the context of the management of this prostate cancer. In this context, a recognized radiological consensus has been established in order to standardize MRI acquisition protocols and the data processing scheme (Prostate Imaging Reporting and Data System, PI-RADS protocol).

Although the improvement provided by multiparametric MRI is significant for the detection of prostate cancer in the clinic, approximately one third of cases remain equivocal. There is therefore a clear clinical advantage in having additional information to support the diagnosis by discriminating between low-grade, intermediate-grade and high-grade tumors and thus reduce the need for biopsies. CEST (chemical exchange saturation transfer) MRI is a promising molecular imaging tool for specifically detecting metabolites containing exchangeable protons present on amide, amine or even hydroxyl functions. MRI-CEST allows non-invasively to highlight molecules of interest such as lactate, glutamate, citrate and other mobile proteins and peptides involved in the carcinogenesis process and usually impossible to visualize by MRI or MRS (Magnetic Resonance Spectroscopy). Exchangeable protons also have the property of seeing their exchange rates modified depending on the surrounding pH, making this CEST contrast sensitive to pH variations. Then, it is APT-CEST (Amide Proton Transfer CEST). The first efforts to translate this method from the preclinical to the clinic were made for brain imaging of gliomas with a significant contribution of APT-CEST in the stratification of tumors. Now, work is expanding to the imaging of other types of tumors such as pelvic tumors, digestive tumors or even breast or lung cancer. Currently, only a few studies have explored CEST MRI in prostate cancer with several limitations both in terms of data acquisition strategy and signal processing. The expertise of the preclinical component of the IVIA platform (In vivo Imaging Auvergne) will make it possible to remove these obstacles and highlight the interest of CEST MRI for the diagnosis and identification of the tumor stage. Thus, the addition of CEST-MRI to the multiparametric MRI strategy will complete the morphological and functional analysis with metabolic criteria that can be decisive in guiding the diagnosis.

The main objective of this study is to study the relationship between the APT-CEST parameter measured in CEST MRI and the gold standard given by the Gleason score (from the anatomopathological analysis of prostate biopsies), these two data being established for each patient.

Secondary objectives are:

* To study the association between all the CEST MRI parameters (APT-CEST, and magnetization transfer ratio with asymmetric analysis (MTRasym) measurements, Guanidyl/APT ratio, Nuclear Overhauser Enhancement (NOE) signal) and:

  * The Gleason score
  * The PI-RADS score, calculated from the readings taken for each of the suspicious lesions identified on multiparametric MRI (T2-weighted anatomical acquisitions and diffusion-weighted DWI or dynamic DCE acquisitions);
  * The measurement of the blood prostate-specific antigen (PSA) level;
  * The volume of the prostate, determined on the anatomical MRI images.
* To situate the predictive potential of CEST measurements in relation to other variables a priori associated with the Gleason score.

DETAILED DESCRIPTION:
This prospective, single-center study will make it possible to evaluate the capabilities of CEST MRI to predict oncological prognosis by comparing it to the reference multiparametric MRI examination and to the anatomopathological analysis of samples taken from biopsies.

When the patient presents a suspicion of prostate cancer identified by an increase in the blood concentration of Prostate Specific Antigen (PSA), he is usually seen in consultation by the urologist within the urology department of the University Hospital. It is during this consultation, after having informed the patient of the need to carry out an MRI to rule out or confirm the presence of a lesion, that the doctor will propose the study to the patient, inform him, and grant him a period of reflection, will answer all his questions and will jointly sign the consent with him if he wishes to participate.

The imaging examination will be carried out a maximum of 6 weeks after the inclusion visit in the research slots of the 3T MRI at CHU Gabriel Montpied (Wednesdays and Fridays). Patients will follow the usual imaging protocol with first multiparametric MRI acquisitions including sequences with injection of contrast product (GADOLINIUM) then a CEST MRI sequence whose duration will not exceed 15 min.

As part of the patient's classic course, if the presence of one or more lesions is proven, a sample of the lesion(s) is taken for an anatomopathological analysis which will give the degree of tumor involvement. The patient returns to the University Hospital approximately 4 weeks later for a consultation for the anatomopathological results and the proposal for subsequent management (monitoring or treatment).

The following data will be noted: age, medical history, PSA level in the blood (nanogram / millilitre), PI-RADS score for each suspicious lesion identified on multiparametric MRI acquisitions, Extension assessment, Parameters measured from the CEST MRI sequence for each of the suspicious lesions: ATP-CEST rate (in arbitrary units), MTRasym, Guanidyl/APT ratio making it possible to assess tumor acidosis, Pathology of samples from the lesion(s): presence or absence of lesions or cancer cells, their number, extent and nature using the Gleason score.

The main objective of this study aims to study the predictive properties of a CEST MRI in the tumor classification of prostate tumors, considering the presence or absence of lesions or cancer cells, their extent and their nature through the score of Gleason on pathological examination of biopsy specimens as dependent variable of interest and measurements on APT-CEST images as main explanatory variable.

False negative rates, diagnostic sensitivity and specificity values and negative and positive predictive values will be presented with a 95% confidence interval.

The concordance between anatomopathological examination and CEST MRI will be studied by estimating the rate of concordant cases and Kappa concordance coefficient.

The usual inferential statistical tests will be considered: for comparisons concerning variables of a quantitative nature: Student's t test or Mann-Whitney test if the conditions for applying the t-test are not respected; for categorical parameters: Chi2 test or Fisher exact test. Particular attention will be paid in particular to the time between the MRI and the pathological examination (3 weeks on average).

ELIGIBILITY:
Inclusion Criteria:

Patients will be included:

* aged over 18
* with suspected prostate cancer identified by an increase in blood PSA concentration
* naïve to chemotherapy, radiotherapy or hormonal therapy
* affiliated to a Social Security system
* able to give informed consent to participate in research
* understanding and reading French well

Exclusion Criteria:

Patients will be excluded:

* refusing to participate in the study
* with impaired understanding, under guardianship/curatorship/deprived of liberty
* presenting "contraindications" to an MRI examination (with administration of a gadolinium chelate): presence of metal parts in the body (electronic devices such as a cardiac pacemaker, a neurostimulator, a cochlear implant, prostheses, intra foreign bodies ocular…), claustrophobia, obesity
* at risk:

  1. . history of allergy to gadolinium (contrast product necessary for performing the multiparmatric MRI planned in the routine care pathway
  2. . history of hypersensitivity to gadoteric acid or gadoline contrast agents, meglumine
* during a period of exclusion from another study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
APT-CEST levels to assess tumoral stage | Measurement at the experimental visit within 3 months after the inclusion visit.
  APT-CEST level is measured on the CEST images and is the maximum, among all the lesions, of the quantitative ratio between the APT-CEST measurement on the area with lesion and the same measurement on the healthy area. The results of the CEST MRI will be collected following the analysis of the metabolic images produced using the tools (Matlab scripts), as well as those developed by the medical image analysis platform (OLEA medical).
Guanidyl/APT ratio to assess tumoral acidosis. | Measurement at the experimental visit within 3 months after the inclusion visit.
  Guanidyl/APT ratio is measured on the CEST images and is the maximum, among all the lesions, of the quantitative ratio between the guanidyl/APT ratio measured on the area with lesion and the same measurement on the healthy area. The results of the CEST MRI will be collected following the analysis of the metabolic images produced using the tools (Matlab scripts), as well as those developed by the medical image analysis platform (OLEA medical).

SECONDARY OUTCOMES:
Gleason score | Measurement at the experimental visit within 3 months after the inclusion visit
  The Gleason score determines the prognosis of prostate cancer based on the architectural structure of the gland. It represent an ordinal score between 2 and 10 depending on the degree of aggressiveness of the cancer.
  * Gleason score 6 (3+3): poorly differentiated and not very aggressive tumors;
  * Gleason score 7 (3+4 or 4+3): moderately differentiated tumors;
  * Gleason score 8, 9 or 10: very undifferentiated and very aggressive tumors.
characterization of highly suspicious lesions on MRI | Measurement at the experimental visit within 3 months after the inclusion visit.
  The PI-RADS (Prostate Imaging Reporting and Data System) score is a prognostic score designed to determine the probability of a cancerous origin of an abnormality visible on MRI. For each abnormality visible on MRI, the radiologist classifies the image according to the Pirads score from the least suspicious (Pirads 1) to the most suspicious (Pirads 5).
Magnetization transfer ratio with asymmetric analysis (MTRasym) complementing the APT-CEST ratio | Measurement at the experimental visit within 3 months after the inclusion visit.
  Quantitative ratios between measurement of the magnetization transfer ratio with asymmetric analysis (MTRasym) on the area with lesion and the healthy area: this measurement will be calculated per lesion and per patient (like the maximum measurements per lesion, on the scale of each patient).
Nuclear Overhauser Enhancement (NOE) measured on CEST-MRI | Measurement at the experimental visit within 3 months after the inclusion visit.
  Quantitative ratios between measurement of the Nuclear Overhauser Enhancement (NOE effect) on the area with lesion and the healthy area: this measurement will be calculated per lesion and per patient (like the maximum measurements per lesion, on the scale of each patient).
Prostate-Specific Antigen PSA level in blood | Measurement at the experimental visit within 3 months after the inclusion visit.
  The prostate-specific antigen (PSA) test is a blood test that can help diagnose prostate problems. The amount of PSA in blood is expressed in nanogram/milliliter. A PSA value of greater than or equal to 4.0 ng/mL is the consensus standard for further prostate cancer evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal CHABROT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, AURA, France